CLINICAL TRIAL: NCT05276245
Title: Testing a New Protocol of Nature-based Intervention to Enhance Well-being: A Randomized Control Trial
Brief Title: Nature-based Intervention to Enhance Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hou Wai Kai, Associate professor, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04465; 2019-2020-0191 (Other: Human Research Ethics Committee)
Record Dates: First submitted 2022-02-22; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Mental Health Wellness 1; Health Behavior; Environmental Exposure
Keywords: nature-based intervention; restorative environments; psychological well-being; health promotion; lunch break
MeSH Terms: conditions — Health Behavior; Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program Group (Experimental): This structured protocol was a 10-day nature-based program with high level of nature engagement and involvement of multiple sensory processes. The program was held in lunch breaks between 12:00 noon and 2:00 p.m. Each session consisted of 30 minutes in the Eco Garden of The Education University of Hong Kong. Activities of this program included walking, ecological photography, sketching butterflies, planting vegetables, drinking herbal tea, observing birds, and taking a nap in nature. Each activity corresponded to specific sensory pathways. For example, butterfly sketching is focused on the use of visual sense, whereas drinking herbal tea involved sense of taste, smell, and touch. Trainers with master's degrees in environmental education and rich experience in guiding ecological tours provided instructions and guidance to participants during the activities. Participants were also asked to pay attention to their surroundings and focus on their five senses during participation.
  Interventions: Behavioral: Structured Protocol of Nature Contact
- Waitlist control group (No Intervention): Participants who were randomly assigned to the waitlist control group were instructed to spend their usual half-hour lunch break in the office for consecutive 10 weekdays. Also, the waitlist control group was told to wait for at least three months before they took part in the structured protocol of nature contact.

INTERVENTIONS:
Behavioral: Structured Protocol of Nature Contact — This structured protocol was a 10-day nature-based program with high level of nature engagement and involvement of multiple sensory processes. The program was held in lunch breaks between 12:00 noon and 2:00 p.m. Each session consisted of 30 minutes in the Eco Garden of The Education University of Hong Kong. Activities of this program included walking, ecological photography, sketching butterflies, planting vegetables, drinking herbal tea, observing birds, and taking a nap in nature. Each activity corresponded to specific sensory pathways. For example, butterfly sketching is focused on the use of visual sense, whereas drinking herbal tea involved sense of taste, smell, and touch. Trainers with master's degrees in environmental education and rich experience in guiding ecological tours provided instructions and guidance to participants during the activities. Participants were also asked to pay attention to their surroundings and focus on their five senses during participation.
  Arms: Program Group

SUMMARY:
The aim of the present study is to investigate the effectiveness of a nature-based intervention on adaptive psychological functioning. We compared a structured protocol with a high level of nature engagement and involvement of multiple sensory processes with a waitlist control group. We expected that participants in the structured protocol of nature contact will report higher levels of mental health and more positive work-related functioning immediately and three months after the interventions.

DETAILED DESCRIPTION:
This study aims to test the associations of nature contact with multiple dimensions of psychological functioning. A total of 90 university employees were randomly assigned to spend their lunch breaks on a (1) 30-minute structured protocol of nature contact and a (2) control group for 10 consecutive weekdays. Psychological distress, psychological well-being, and work-related psychological outcomes were assessed at baseline (T1), the day after the 10-day intervention (T2), and three months after the intervention (T3).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Cantonese speaking
* Full-time employment of The Education University of Hong Kong

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline (T1) anxiety symptoms to post intervention (T2) and follow up (T3) | Before the intervention (T1), the day after the 10-day intervention (T2), and three months after the intervention (T3).
  The Chinese version of the 7-item Generalized Anxiety Disorder (GAD-7) was used to measure anxiety symptoms at all time points. Participants rated each item on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day) based on their experience in the past two weeks. Higher scores indicated greater severity of anxiety symptoms (range = 0-21).
Change from baseline (T1) depressive symptoms to post intervention (T2) and follow up (T3) | Before the intervention (T1), the day after the 10-day intervention (T2), and three months after the intervention (T3).
  Depressive symptoms were measured using the Chinese version of the Patient Health Questionnaire-9 (PHQ-9) at T1, T2, and T3, respectively. Participants rated each item on a 4-point scale as in GAD-7. Higher scores indicate the greatest severity of the depressive symptoms (range 0-27).
Change from baseline (T1) perceived stress to post intervention (T2) and follow up (T3) | Before the intervention (T1), the day after the 10-day intervention (T2), and three months after the intervention (T3).
  Perceived stress was assessed at all time points using the Chinese version of the 10-item Perceived Stress Scale (PSS-10). Participants reported their subjective stress in the past two weeks on a 5-point scale (0 = never, 4 = very often). Total scores ranged from 0 to 40, with higher scores indicating higher levels of perceived stress.
Change from baseline (T1) subjective well-being to post intervention (T2) and follow up (T3) | Before the intervention (T1), the day after the 10-day intervention (T2), and three months after the intervention (T3).
  The WHO-Five Well-being Index (WHO-5) consisted of five positively worded items. Participants were asked to report the presence of the five positive mental states in the past 2 weeks on a 6-point scale ranging from 0 (at no time) to 5 (all of the time).
Change from baseline (T1) satisfaction with life to post intervention (T2) and follow up (T3) | Before the intervention (T1), the day after the 10-day intervention (T2), and three months after the intervention (T3).
  Satisfaction with Life Scale (SWLS) was used to assess participants' well-being with regard to satisfaction and fulfillment of their current state on a 4-point scale (1 = strongly disagree, 4 = strongly agree). The five items were summed, with higher scores indicating higher life satisfaction (range = 5-20).
Change from baseline (T1) positive affect to post intervention (T2) and follow up (T3) | Before the intervention (T1), the day after the 10-day intervention (T2), and three months after the intervention (T3).
  The 10-item positive affect subscale of Chinese Affect Scale (CAS-PA) assessed frequency of positive emotional experience in the past 2 weeks on a 5-point scale (0 = not at all, 4 = all the time).
Change from baseline (T1) burnout to post intervention (T2) and follow up (T3) | Before the intervention (T1), the day after the 10-day intervention (T2), and three months after the intervention (T3).
  Burnout was measured using the Chinese version of the 14-item Maslach Burnout Inventory-General Survey (MBI-GS) at all time points. Participants rated how often they had different experiences of burnout in the past two weeks on a 7-point scale (0 = never, 6 = always). The scale consisted of five questions on emotional exhaustion, four on cynicism, and five on professional efficacy.
Change from baseline (T1) work engagement to post intervention (T2) and follow up (T3) | Before the intervention (T1), the day after the 10-day intervention (T2), and three months after the intervention (T3).
  The Chinese version of the 17-item Utrecht Work Engagement Scale (UWES) was used to assess vigor, dedication, and absorption at work at all time points. Participants indicated the frequency of these experiences at work in the past two weeks on a 7-point scale (0 = never, 6 = always).

CONTACTS AND LOCATIONS:
Overall Officials: Wai Kai Hou, PhD, Principal Investigator — The Education University of Hong Kong
Locations (1):
- The Education University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be available on request.